CLINICAL TRIAL: NCT02033889
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, 26-Week Multicenter Study With a 78-Week Extension To Evaluate The Efficacy And Safety Of Ertugliflozin In Subjects With Type 2 Diabetes Mellitus And Inadequate Glycemic Control On Metformin Monotherapy.
Brief Title: A Study To Evaluate The Efficacy And Safety Of Ertugliflozin In Participants With Type 2 Diabetes Mellitus And Inadequate Glycemic Control On Metformin Monotherapy (MK-8835-007).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8835-007; 2013-003290-95 (EudraCT Number); B1521017 (Other: Pfizer Protocol Number); MK-8835-007 (Other: Merck Protocol Number)
Record Dates: First submitted 2014-01-09; First posted 2014-01-13 (Estimated); Results first posted 2018-09-10 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ertugliflozin; glimepiride; Insulin Glargine; Insulin Detemir; Insulin, Isophane; insulin degludec; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ertuglifozin 5 mg (Experimental): Ertugliflozin 5 mg orally, once daily from Day 1 to Week 104. Up to 26 weeks, participants meeting glycemic rescue criteria were rescued with open-label glimepiride, and if they met rescue criteria again, and they were on maximal tolerated doses of glimepiride, they received basal insulin. After Week 26, non-rescued participants who had a fasting finger-stick glucose ≥110 mg/dL received glimepiride/placebo. If a participant met glycemic rescue criteria after 26 weeks, and they were on maximal tolerated dose of glimepiride, then rescue with basal insulin was initiated.
  Interventions: Drug: Ertugliflozin 5 mg; Drug: Placebo to Ertugliflozin; Other: Glimepiride; Drug: Placebo to Glimepiride; Biological: Basal Insulin; Drug: Metformin
- Ertugliflozin 15 mg (Experimental): Ertugliflozin 15 mg orally, once daily from Day 1 to Week 104. Up to 26 weeks, participants meeting glycemic rescue criteria were rescued with open-label glimepiride, and if they met rescue criteria again, and they were on maximal tolerated doses of glimepiride, they received basal insulin. After Week 26, non-rescued participants who had a fasting finger-stick glucose ≥110 mg/dL received glimepiride/placebo. If a participant met glycemic rescue criteria after 26 weeks, and they were on maximal tolerated dose of glimepiride, then rescue with basal insulin was initiated.
  Interventions: Drug: Ertugliflozin 15 mg; Other: Glimepiride; Drug: Placebo to Glimepiride; Biological: Basal Insulin; Drug: Metformin
- Placebo/Glimepiride (Placebo Comparator): Placebo to ertugliflozin, orally once daily from Day 1 to Week 104. Up to 26 weeks, participants meeting glycemic rescue criteria were rescued with open-label glimepiride, and if they met rescue criteria again, and they were on maximal tolerated doses of glimepiride, they received basal insulin. After Week 26, non-rescued participants who had a fasting finger-stick glucose ≥110 mg/dL received blinded glimepiride. If a participant met glycemic rescue criteria after 26 weeks, and they were on maximal tolerated dose of glimepiride, then rescue with basal insulin was initiated.
  Interventions: Drug: Placebo to Ertugliflozin; Other: Glimepiride; Biological: Basal Insulin; Drug: Metformin

INTERVENTIONS:
Drug: Ertugliflozin 5 mg — Ertugliflozin 5 mg orally (1 ertugliflozin 5 mg tablet and 1 placebo ertugliflozin 10 mg tablet), once daily from Day 1 to Week 104.
  Other Names: MK-8835
  Arms: Ertuglifozin 5 mg
Drug: Ertugliflozin 15 mg — Ertugliflozin 15 mg orally (1 ertugliflozin 5 mg tablet and 1 ertugliflozin 10 mg tablet), once daily from Day 1 to Week 104.
  Other Names: MK-8835
  Arms: Ertugliflozin 15 mg
Drug: Placebo to Ertugliflozin — Placebo to ertuglioflozin (1 placebo ertugliflozin 5 mg tablet and/or 1 placebo ertugliflozin 10 mg tablet), orally once daily from Day 1 to Week 104.
  Arms: Ertuglifozin 5 mg; Placebo/Glimepiride
Other: Glimepiride — Open-label Glimepiride will be used for glycemic rescue therapy (up to a maximum of 6 or 8 mg per day, based on the local label of glimepiride) in the 26-week initial period. Blinded Glimepiride (up to a maximum of 6 or 8 mg per day, based on the local label of glimepiride will be used in the 78-week extension period in participants who were not rescued with open-label glimepiride during the 26-week initial period.
  Other Names: Amaryl; GLIMPID; GLIMY
Drug: Placebo to Glimepiride — Placebo to glimepiride will be used in the 78-week extension period in participants who were not rescued with open-label glimepiride during the 26-week initial period. Dosing and titration of placebo to glimepiride is at the discretion of the investigator.
  Arms: Ertugliflozin 15 mg; Ertuglifozin 5 mg
Biological: Basal Insulin — Basal insulin will be administered in the initial 26-week period for participants with glucose values exceeding protocol-specified values and for participants requiring rescue therapy in the 78-week extension period. Dosing and titration of basal insulin is at the discretion of the Investigator.
  Other Names: Insulin glargine; Insulin detemir; NPH insulin; Degludec
Drug: Metformin — Metformin >=1500 mg/day, orally, once a day
  Other Names: Glucophage XR; Carbophage SR; Riomet; Fortamet; Glumetza; Obimet; Gluformin; Dianben; Diabex; Diaformin; Siofor; Metfogamma

SUMMARY:
This is an efficacy and safety study of ertugliflozin in participants with type 2 diabetes mellitus (T2DM) and inadequate glycemic control on metformin monotherapy. The primary study hypothesis is that at Week 26, the mean reduction from baseline in hemoglobin A1c (HbA1c) for ertugliflozin is greater than that for placebo.

DETAILED DESCRIPTION:
The trial includes a 13-15 week run-in period prior to randomization, and a 26-week, double-blind, placebo-controlled treatment period followed by a 78-week double-blind, extension period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T2DM in accordance to American Diabetes Association guidelines
* Participants must be receiving metformin monotherapy for less than 8 weeks prior to study participation or require change in their diabetes regimen to remain eligible to participate in the trial (including discontinuing anti-hyperglycemic agent [AHA] therapy) and must have a hemoglobin A1c of 7.0 to 10.5% (53-91 mmol/mol) after at least 8 weeks on a regimen of metformin monotherapy

Exclusion Criteria:

* History of myocardial infarction, unstable angina, arterial revascularization, stroke, transient ischemic attack, or New York Heart Association (NYHA) functional class III-IV heart failure within 3 months of study participation
* A clinically significant electrocardiogram abnormality
* A history of malignancy ≤5 years prior to study participation, except for adequately treated basal or squamous cell skin cancer or in situ cervical cancer
* A known hypersensitivity or intolerance to any sodium-glucose co-transporter 2 (SGLT2) inhibitor or glimepiride
* On a blood pressure or lipid altering medication that have not been on a stable dose for at least 4 weeks prior to study participation
* A surgical procedure within 6 weeks prior to study participation or planned major surgery during the trial
* Donation of blood or blood products within 6 weeks of study participation or plans to donate blood or blood products at any time during the trial
* Pregnant or breast-feeding, or is expecting to conceive during the trial, including 14 days following the last dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 621 (Actual)
Dates: Start 2013-12-13 (Actual); Primary Completion 2017-08-03 (Actual); Study Completion 2017-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Rosenstock J, Frias J, Pall D, Charbonnel B, Pascu R, Saur D, Darekar A, Huyck S, Shi H, Lauring B, Terra SG. Effect of ertugliflozin on glucose control, body weight, blood pressure and bone density in type 2 diabetes mellitus inadequately controlled on metformin monotherapy (VERTIS MET). Diabetes Obes Metab. 2018 Mar;20(3):520-529. doi: 10.1111/dom.13103. Epub 2017 Oct 2. PMID 28857451
- [Derived] Ji L, Liu J, Xu ZJ, Wei Z, Zhang R, Malkani S, Cater NB, Frederich R. Efficacy and Safety of Ertugliflozin Added to Metformin: A Pooled Population from Asia with Type 2 Diabetes and Overweight or Obesity. Diabetes Ther. 2023 Feb;14(2):319-334. doi: 10.1007/s13300-022-01345-6. Epub 2023 Feb 3. PMID 36763328
- [Derived] Fediuk DJ, Sahasrabudhe V, Dawra VK, Zhou S, Sweeney K. Population Pharmacokinetic Analyses of Ertugliflozin in Select Ethnic Populations. Clin Pharmacol Drug Dev. 2021 Nov;10(11):1297-1306. doi: 10.1002/cpdd.970. Epub 2021 Jul 2. PMID 34213819
- [Derived] Gallo S, Calle RA, Terra SG, Pong A, Tarasenko L, Raji A. Effects of Ertugliflozin on Liver Enzymes in Patients with Type 2 Diabetes: A Post-Hoc Pooled Analysis of Phase 3 Trials. Diabetes Ther. 2020 Aug;11(8):1849-1860. doi: 10.1007/s13300-020-00867-1. Epub 2020 Jul 9. PMID 32648108
- [Derived] Patel S, Hickman A, Frederich R, Johnson S, Huyck S, Mancuso JP, Gantz I, Terra SG. Safety of Ertugliflozin in Patients with Type 2 Diabetes Mellitus: Pooled Analysis of Seven Phase 3 Randomized Controlled Trials. Diabetes Ther. 2020 Jun;11(6):1347-1367. doi: 10.1007/s13300-020-00803-3. Epub 2020 May 5. PMID 32372382
- [Derived] Liu J, Tarasenko L, Pong A, Huyck S, Wu L, Patel S, Hickman A, Mancuso JP, Gantz I, Terra SG. Efficacy and safety of ertugliflozin across racial groups in patients with type 2 diabetes mellitus. Curr Med Res Opin. 2020 Aug;36(8):1277-1284. doi: 10.1080/03007995.2020.1760228. Epub 2020 May 13. PMID 32324082
- [Derived] Liu J, Tarasenko L, Pong A, Huyck S, Patel S, Hickman A, Mancuso JP, Ellison MC, Gantz I, Terra SG. Efficacy and safety of ertugliflozin in Hispanic/Latino patients with type 2 diabetes mellitus. Curr Med Res Opin. 2020 Jul;36(7):1097-1106. doi: 10.1080/03007995.2020.1760227. Epub 2020 May 13. PMID 32324065
- [Derived] Cherney DZI, Heerspink HJL, Frederich R, Maldonado M, Liu J, Pong A, Xu ZJ, Patel S, Hickman A, Mancuso JP, Gantz I, Terra SG. Effects of ertugliflozin on renal function over 104 weeks of treatment: a post hoc analysis of two randomised controlled trials. Diabetologia. 2020 Jun;63(6):1128-1140. doi: 10.1007/s00125-020-05133-4. Epub 2020 Mar 31. PMID 32236732
- [Derived] Liu J, Patel S, Cater NB, Wu L, Huyck S, Terra SG, Hickman A, Darekar A, Pong A, Gantz I. Efficacy and safety of ertugliflozin in East/Southeast Asian patients with type 2 diabetes mellitus. Diabetes Obes Metab. 2020 Apr;22(4):574-582. doi: 10.1111/dom.13931. Epub 2020 Jan 3. PMID 31797522
- [Derived] Liu J, Pong A, Gallo S, Darekar A, Terra SG. Effect of ertugliflozin on blood pressure in patients with type 2 diabetes mellitus: a post hoc pooled analysis of randomized controlled trials. Cardiovasc Diabetol. 2019 May 7;18(1):59. doi: 10.1186/s12933-019-0856-7. PMID 31064361
- [Derived] Gallo S, Charbonnel B, Goldman A, Shi H, Huyck S, Darekar A, Lauring B, Terra SG. Long-term efficacy and safety of ertugliflozin in patients with type 2 diabetes mellitus inadequately controlled with metformin monotherapy: 104-week VERTIS MET trial. Diabetes Obes Metab. 2019 Apr;21(4):1027-1036. doi: 10.1111/dom.13631. Epub 2019 Feb 14. PMID 30614616

RESULTS

PARTICIPANT FLOW:
Groups:
- Ertugliflozin 5 mg: Ertugliflozin 5 mg orally, once daily from Day 1 to Week 104. Up to 26 weeks, participants meeting glycemic rescue criteria were rescued with open-label glimepiride, and if they met rescue criteria again, and they were on maximal tolerated doses of glimepiride, they received basal insulin. After Week 26, non-rescued participants who had a fasting finger-stick glucose ≥110 mg/dL received glimepiride/placebo. If a participant met glycemic rescue criteria after 26 weeks, and they were on maximal tolerated dose of glimepiride, then rescue with basal insulin was initiated.
Period: Overall Study
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Started | 209 | 207 | 205
Completed | 175 | 187 | 180
Not Completed | 34 | 20 | 25
Not completed — Adverse Event | 3 | 1 | 3
Not completed — Death | 3 | 1 | 2
Not completed — Excluded Medication | 1 | 1 | 0
Not completed — Lost to Follow-up | 8 | 5 | 6
Not completed — Non-Compliance With Study Drug | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 1
Not completed — Participant moved | 0 | 1 | 0
Not completed — Withdrawal by Subject | 18 | 10 | 13

BASELINE CHARACTERISTICS:
Population: All randomized and treated participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Total
Number analyzed (Participants) | 209 | 207 | 205 | 621
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: All randomized and treated participants
  Years | 56.5 (8.7) | 56.6 (8.2) | 56.9 (9.4) | 56.6 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All randomized and treated participants
  Participants
    Female | 111 | 110 | 112 | 333
    Male | 98 | 97 | 93 | 288
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: All randomized and treated participants
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 31 | 34 | 35 | 100
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 19 | 22 | 23 | 64
    White | 144 | 134 | 133 | 411
    More than one race | 15 | 17 | 14 | 46
    Unknown or Not Reported | 0 | 0 | 0 | 0
Baseline Hemoglobin A1C (A1C) [Mean (Standard Deviation); unit: Percentage A1C] — Percentage A1C is the ratio of glycated hemoglobin to total hemoglobin x 100. Population: All randomized participants who have received at least one dose of investigational product and have a measurement of baseline A1C.
  Percentage A1C
    number analyzed (Participants) | 207 | 205 | 202 | 614
    (all) | 8.17 (0.90) | 8.06 (0.89) | 8.13 (0.93) | 8.12 (0.90)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] — Population: All randomized participants who have received at least one dose of investigational product and have a measurement of baseline FPG.
  mg/dL
    number analyzed (Participants) | 202 | 199 | 203 | 604
    (all) | 169.1 (41.7) | 168.1 (45.5) | 167.5 (44.4) | 168.3 (43.8)
Body Weight [Mean (Standard Deviation); unit: Kilograms] — Population: All randomized and treated participants who had a baseline Body Weight.
  Kilograms | 84.5 (17.1) | 84.8 (17.2) | 85.3 (16.5) | 84.9 (16.9)
Sitting Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: mmHg] — Population: All randomized participants who have received at least one dose of investigational product and have a measurement of baseline SBP.
  mmHg
    number analyzed (Participants) | 201 | 201 | 198 | 600
    (all) | 129.30 (15.43) | 130.48 (13.77) | 130.37 (12.00) | 130.05 (13.80)
Diastolic Blood Pressure (DBP) [Mean (Standard Deviation); unit: mmHg] — Population: All randomized participants who have received at least one dose of investigational product and have a measurement of baseline DBP.
  mmHg
    number analyzed (Participants) | 201 | 201 | 198 | 600
    (all) | 77.45 (7.55) | 78.45 (8.32) | 78.08 (7.45) | 77.99 (7.78)
Bone Mineral Density (BMD) as Measured by Dual Energy X-Ray Absorptiometry (DXA) of the Femoral Neck [Mean (Standard Deviation); unit: g/cm^2] — BMD at the femoral neck was assessed by DXA at baseline. Population: All randomized participants who have received at least one dose of investigational product and have a measurement of baseline BMD of the femoral neck.
  g/cm^2 | 0.92 (0.17) | 0.92 (0.16) | 0.89 (0.15) | 0.91 (0.16)
BMD as Measured by DXA of the Lumbar Spine (L1-L4) [Mean (Standard Deviation); unit: g/cm^2] — BMD at the lumbar spine (L1-L4) was assessed by DXA at baseline. Population: All randomized participants who have received at least one dose of investigational product and have a measurement of baseline BMD of the lumbar spine (L1-L4).
  g/cm^2
    number analyzed (Participants) | 209 | 207 | 204 | 620
    (all) | 1.15 (0.18) | 1.13 (0.18) | 1.10 (0.17) | 1.13 (0.18)
BMD as Measured by DXA of the Total hip [Mean (Standard Deviation); unit: g/cm^2] — BMD at the total hip was assessed by DXA at baseline. Population: All randomized participants who have received at least one dose of investigational product and have a measurement of baseline BMD of the total hip.
  g/cm^2 | 1.06 (0.15) | 1.07 (0.15) | 1.04 (0.14) | 1.06 (0.15)
BMD as Measured by DXA at the Distal Forearm [Mean (Standard Deviation); unit: g/cm^2] — BMD at the distal forearm was assessed by DXA at baseline. Population: All randomized participants who have received at least one dose of investigational product and have a measurement of baseline BMD of the distal forearm.
  g/cm^2
    number analyzed (Participants) | 209 | 205 | 205 | 619
    (all) | 0.81 (0.14) | 0.81 (0.14) | 0.79 (0.13) | 0.80 (0.14)
Bone Biomarker Carboxy-Terminal Cross-Linking Telopeptides of Type I Collagen (CTX) [Mean (Standard Deviation); unit: ng/L] — CTX is a biochemical marker of bone resorption. Population: All randomized participants who have received at least one dose of investigational product and have a measurement of baseline CTX.
  ng/L
    number analyzed (Participants) | 200 | 196 | 195 | 591
    (all) | 268.3 (132.9) | 266.9 (129.9) | 273.0 (135.2) | 269.4 (132.5)
Bone Biomarker Procollagen Type I N-terminal Propeptide (P1NP) [Mean (Standard Deviation); unit: microgm/L] — P1NP is a biochemical marker of bone resorption. Population: All randomized participants who have received at least one dose of investigational product and have a measurement of baseline P1NP.
  microgm/L
    number analyzed (Participants) | 200 | 198 | 198 | 596
    (all) | 32.0 (15.0) | 32.8 (14.5) | 31.6 (16.5) | 32.1 (15.3)
Bone Biomarker Parathyroid Hormone (PTH) [Mean (Standard Deviation); unit: ng/L] — PTH is a biochemical marker of bone resorption. Population: All randomized participants who have received at least one dose of investigational product and have a measurement of baseline PTH.
  ng/L
    number analyzed (Participants) | 202 | 194 | 200 | 596
    (all) | 19.29 (8.17) | 19.52 (6.91) | 19.97 (7.73) | 19.59 (7.62)
Menopausal Status [Count of Participants; unit: Participants] — Menopausal status includes men, premenopausal women, women who are perimenopausal or <3 years postmenopausal, women who are ≥3 years postmenopausal. Population: All randomized participants who have received at least one dose of investigational product and have menopausal status baseline information.
  Participants
    Male | 98 | 97 | 93 | 288
    Premenopausal Women | 16 | 17 | 16 | 49
    Perimenopausal or <3 yrs. postmen. | 9 | 10 | 11 | 30
    Women ≥3 years postmenopausal | 86 | 83 | 85 | 254
Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73 m^2] — Population: All randomized participants who have received at least one dose of investigational product and have a measurement of baseline eGFR.
  mL/min/1.73 m^2 | 91.6 (19.8) | 88.9 (17.5) | 91.1 (20.6) | 90.5 (19.3)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in A1C at Week 26 (Excluding Rescue Approach)
Description: A1C is blood marker used to report average blood glucose levels over prolonged periods of time. Percentage A1C is the ratio of glycated hemoglobin to total hemoglobin x 100. Thus, this change from baseline reflects the Week 26 A1C minus the Week 0 A1C (which is estimated on average for each treatment group using a constrained longitudinal data analysis model, which allows for participants with missing data to be included in the analysis). Participants who met pre-specified glycemic criteria were rescued with oral tablets of open-label glimepiride or basal insulin injected subcutaneously, and dosed according to Investigator judgment. Per protocol, this data set excludes data for any participant after the initiation of glycemic rescue therapy.
Time Frame: Baseline and Week 26
Population: All randomized participants who took at least one dose of study medication and had at least one assessment of the respective endpoint at baseline or post-baseline up to Week 26.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent A1C
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 209 | 207 | 205
Percent A1C | -0.03 [-0.15 to 0.10] | -0.73 [-0.85 to -0.61] | -0.91 [-1.03 to -0.78]
Statistical Analysis 1: Comparison: Placebo/Glimepiride vs Ertugliflozin 15 mg; Test type: Superiority; p < 0.001, Constrained Longitudinal Data Analysis; Difference in Least Squares Means = -0.88, 95% CI 2-sided [-1.05 to -0.71]; Based on Constrained Longitudinal Data Analysis (cLDA) model with fixed effects for treatment, time, prior anti hyperglycemic medication (Metformin monotherapy or Metformin + another anti-hyperglycemic agent, AHA), baseline eGFR (continuous), menopausal status. Time was treated as a categorical variable
Statistical Analysis 2: Comparison: Placebo/Glimepiride vs Ertugliflozin 5 mg; Test type: Superiority; p < 0.001, Constrained Longitudinal Data Analysis; Difference in Least Squares Means = -0.70, 95% CI 2-sided [-0.87 to -0.53]; Based on cLDA model with fixed effects for treatment, time, prior anti hyperglycemic medication (Metformin monotherapy or Metformin + another anti-hyperglycemic agent, AHA), baseline eGFR (continuous), menopausal status. Time was treated as a categorical variable

2. Primary Outcome: Percentage of Participants Experiencing An Adverse Event (AE) (Including Rescue Approach)
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. Per protocol, participants who met pre-specified glycemic criteria were rescued with open-label glimepiride or basal insulin according to Investigator judgment.
Time Frame: Up to Week 106
Population: All participants who received at least one dose of investigational product.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 209 | 207 | 205
Percentage of Participants | 77.5 | 70.5 | 75.6

3. Primary Outcome: Percentage of Participants Discontinuing Study Treatment Due to an AE (Including Rescue Approach)
Description: as for outcome 2
Time Frame: Up to Week 104
Population: All participants who received at least one dose of investigational product.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 209 | 207 | 205
Percentage of Participants | 2.4 | 3.4 | 3.9
Statistical Analysis 1: Comparison: Placebo/Glimepiride vs Ertugliflozin 15 mg; Test type: Other; Difference in % vs Placebo/Glimepiride = 1.5, 95% CI 2-sided [-2.1 to 5.4]; Miettinen & Nurminen method was used to construct the 95% CI
Statistical Analysis 2: Comparison: Placebo/Glimepiride vs Ertugliflozin 5 mg; Test type: Other; Difference in % vs Placebo/Glimepiride = 1.0, 95% CI 2-sided [-2.5 to 4.7]; Miettinen & Nurminen method was used to construct the 95% CI

4. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 26 (Excluding Rescue Approach)
Description: Blood glucose was measured on a fasting basis. Blood was drawn at predose on Day 1 and after 26 weeks of treatment to determine change in plasma glucose levels (i.e., FPG at Week 26 minus FPG at Week 0) which is estimated on average for each treatment group using a constrained longitudinal data analysis model, which allows for participants with missing data to be included in the analysis. Participants who met pre-specified glycemic criteria were rescued with oral tablets of open-label glimepiride or basal insulin injected subcutaneously, and dosed according to Investigator judgment. Per protocol, this data set excludes data for any participant after the initiation of glycemic rescue therapy.
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 209 | 207 | 205
mg/dL | -0.85 [-5.93 to 4.23] | -27.54 [-32.36 to -22.73] | -39.10 [-43.96 to -34.23]
Statistical Analysis 1: Comparison: Placebo/Glimepiride vs Ertugliflozin 15 mg; Test type: Superiority; p < 0.001, Constrained Longitudinal Data Analysis; Difference in Least Squares Means = -38.25, 95% CI 2-sided [-44.50 to -31.99]; Based on the cLDA model with fixed effects for treatment, time, prior antihyperglycemic medication (metformin monotherapy or metformin + another AHA), baseline eGFR (continuous), menopausal status. Time was treated as a categorical variable
Statistical Analysis 2: Comparison: Placebo/Glimepiride vs Ertugliflozin 5 mg; Test type: Superiority; p < 0.001, Constrained Longitudinal Data Analysis; Difference in the Least Squares Means = -26.69, 95% CI 2-sided [-32.90 to -20.48]; [other analysis details as in outcome 4, analysis 1]

5. Secondary Outcome: Change From Baseline in Body Weight at Week 26 (Excluding Rescue Approach)
Description: The change in body weight from baseline reflects the Week 26 body weight minus the Week 0 body weight (which is estimated on average for each treatment group using a constrained longitudinal data analysis model, which allows for participants with missing data to be included in the analysis). Participants who met pre-specified glycemic criteria were rescued with oral tablets of open-label glimepiride or basal insulin injected subcutaneously, and dosed according to Investigator judgment. Per protocol, this data set excludes data for any participant after the initiation of glycemic rescue therapy.
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Kilograms
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 209 | 207 | 205
Kilograms | -1.33 [-1.74 to -0.92] | -3.01 [-3.40 to -2.62] | -2.93 [-3.33 to -2.53]
Statistical Analysis 1: Comparison: Placebo/Glimepiride vs Ertugliflozin 15 mg; Test type: Superiority; p < 0.001, Constrained Longitudinal Data Analysis; Difference in Least Squares Means = -1.60, 95% CI 2-sided [-2.16 to -1.03]; [other analysis details as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Placebo/Glimepiride vs Ertugliflozin 5 mg; Test type: Superiority; p < 0.001, Constrained Longitudinal Data Analysis; Difference in Least Squares Means = -1.67, 95% CI 2-sided [-2.24 to -1.11]; [other analysis details as in outcome 4, analysis 1]

6. Secondary Outcome: Percentage of Participants With an A1C of <7% (53 mmol/Mol) at Week 26 (Logistic Regression Using Multiple Imputation: Excluding Rescue Approach)
Description: A1C is blood marker used to report average blood glucose levels over prolonged periods of time and is reported as a percentage (%). Percentage A1C is the ratio of glycated hemoglobin to total hemoglobin x 100. Participants who met pre-specified glycemic criteria were rescued with oral tablets of open-label glimepiride or basal insulin injected subcutaneously, and dosed according to Investigator judgment. Per protocol, this data set excludes data for any participant after the initiation of glycemic rescue therapy.
Time Frame: Week 26
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 209 | 207 | 205
Percentage of Participants | 15.8 | 35.3 | 40.0
Statistical Analysis 1: Comparison: Placebo/Glimepiride vs Ertugliflozin 15 mg; Test type: Superiority; p < 0.001, Regression, Logistic; Adjusted Odds Ratio Relative to Placebo = 4.48, 95% CI 2-sided [2.64 to 7.62]; Adjusted odds ratio based on a logistic regression model fitted with fixed effects for treatment, prior antihyperglycemic medication (metformin monotherapy or metformin + another AHA), menopausal status, covariates for baseline A1C and baseline eGFR (continuous). Missing data imputed using a multiple imputation procedure based on cLDA prediction modeling with fixed effects as in the primary analysis, which allows for participants with missing data to be included in the analysis
Statistical Analysis 2: Comparison: Placebo/Glimepiride vs Ertugliflozin 5 mg; Test type: Superiority; p < 0.001, Regression, Logistic; Adjusted Odds Ratio Relative to Placebo = 3.03, 95% CI 2-sided [1.81 to 5.06]; [other analysis details as in outcome 6, analysis 1]

7. Secondary Outcome: Change From Baseline in Sitting Systolic Blood Pressure at Week 26 (Excluding Rescue Approach)
Description: This change from baseline reflects the Week 26 sitting systolic blood pressure (SBP) minus the Week 0 sitting SBP (which is estimated on average for each treatment group using a constrained longitudinal data analysis model, which allows for participants with missing data to be included in the analysis). Participants who met pre-specified glycemic criteria were rescued with oral tablets of open-label glimepiride or basal insulin injected subcutaneously, and dosed according to Investigator judgment. Per protocol, this data set excludes data for any participant after the initiation of glycemic rescue therapy.
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 209 | 207 | 204
mmHg | -0.70 [-2.46 to 1.06] | -4.38 [-6.01 to -2.75] | -5.20 [-6.87 to -3.54]
Statistical Analysis 1: Comparison: Placebo/Glimepiride vs Ertugliflozin 15 mg; Test type: Superiority; p < 0.001, Constrained Longitudinal Data Analysis; Difference in Least Squares Means = -4.50, 95% CI 2-sided [-6.81 to -2.19]; Based on the cLDA model with fixed effects for treatment, time, prior antihyperglycemic medication (metformin monotherapy or metformin + another AHA), baseline eGFR (continuous), menopausal status, and the interaction of time by treatment. Time was treated as a categorical variable
Statistical Analysis 2: Comparison: Placebo/Glimepiride vs Ertugliflozin 5 mg; Test type: Superiority; p = 0.002, Constrained Longitudinal Data Analysis; Difference in Least Squares Means = -3.68, 95% CI 2-sided [-5.96 to -1.39]; [other analysis details as in outcome 7, analysis 1]

8. Secondary Outcome: Change From Baseline in Sitting Diastolic Blood Pressure at Week 26 (Excluding Rescue Approach)
Description: This change from baseline reflects the Week 26 sitting diastolic blood pressure (DBP) minus the Week 0 sitting DBP (which is estimated on average for each treatment group using a constrained longitudinal data analysis model, which allows for participants with missing data to be included in the analysis). Participants who met pre-specified glycemic criteria were rescued with oral tablets of open-label glimepiride or basal insulin injected subcutaneously, and dosed according to Investigator judgment. Per protocol, this data set excludes data for any participant after the initiation of glycemic rescue therapy.
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 209 | 207 | 204
mmHg | 0.23 [-0.85 to 1.31] | -1.59 [-2.59 to -0.59] | -2.19 [-3.21 to -1.17]
Statistical Analysis 1: Comparison: Placebo/Glimepiride vs Ertugliflozin 15 mg; Test type: Superiority; p = 0.001, Constrained Longitudinal Data Analysis; Difference in Least Squares Means = -2.42, 95% CI 2-sided [-3.86 to -0.98]; [other analysis details as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Placebo/Glimepiride vs Ertugliflozin 5 mg; Test type: Superiority; p = 0.013, Constrained Longitudinal Data Analysis; Difference in Least Squares Means = -1.82, 95% CI 2-sided [-3.24 to -0.39]; [other analysis details as in outcome 7, analysis 1]

9. Secondary Outcome: Percentage of Participants With an A1C of <6.5% (48 mmol/Mol) at Week 26 (Logistic Regression Using Multiple Imputation: Excluding Rescue Approach)
Description: as for outcome 6
Time Frame: Week 26
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 209 | 207 | 205
Percentage of Participants | 2.9 | 8.7 | 12.2
Statistical Analysis 1: Comparison: Placebo/Glimepiride vs Ertugliflozin 15 mg; Test type: Superiority; p < 0.001, Regression, Logistic; Adjusted Odds Ratio = 5.41, 95% CI 2-sided [2.10 to 13.90]; [other analysis details as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Placebo/Glimepiride vs Ertugliflozin 5 mg; Test type: Superiority; p = 0.023, Regression, Logistic; Adjusted Odds Ratio = 3.10, 95% CI 2-sided [1.17 to 8.22]; [other analysis details as in outcome 6, analysis 1]

10. Secondary Outcome: Percentage of Participants Receiving Glycemic Rescue Therapy up to Week 26
Description: Per protocol, participants who met pre-specified glycemic criteria were rescued with oral tablets of open-label glimepiride or basal insulin injected subcutaneously, and dosed according to Investigator judgment.
Time Frame: Up to Week 26
Population: All participants who received at least one dose of investigational product.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 209 | 207 | 205
Percentage of Participants | 17.7 | 2.9 | 1.5
Statistical Analysis 1: Comparison: Placebo/Glimepiride vs Ertugliflozin 15 mg; Test type: Superiority; p < 0.001, Miettinen & Nurminen method; Miettinen & Nurminen method was used to construct both the 95% CI and derive p-value for the difference between the proportions (i.e. percentages); Difference in % vs Placebo = -16.2, 95% CI 2-sided [-22.2 to -11.2]
Statistical Analysis 2: Comparison: Placebo/Glimepiride vs Ertugliflozin 5 mg; Test type: Superiority; p < 0.001, Miettinen & Nurminen method; [statistical method as in outcome 10, analysis 1]; Difference in % vs Placebo = -14.8, 95% CI 2-sided [-20.9 to -9.4]

11. Secondary Outcome: Time to Glycemic Rescue Therapy at Week 26
Description: as for outcome 10
Time Frame: Week 26
Population: All participants who received at least one dose of investigational product and received glycemic rescue through Week 26.
Measure: Median (Full Range); unit: Days
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 36 | 6 | 3
Days | 105 [15 to 183] | 112 [23 to 151] | 139 [127 to 145]

12. Secondary Outcome: Change From Baseline in A1C at Week 52 (Excluding Rescue Approach)
Description: A1C is blood marker used to report average blood glucose levels over prolonged periods of time. Percentage A1C is the ratio of glycated hemoglobin to total hemoglobin x 100. Thus, this change from baseline reflects the Week 52 A1C minus the Week 0 A1C. Participants who met pre-specified glycemic criteria were rescued with oral tablets of open-label glimepiride or basal insulin injected subcutaneously, and dosed according to Investigator judgment. Per protocol, this data set excludes data for any participant after the initiation of glycemic rescue therapy.
Time Frame: Baseline and Week 52
Population: All randomized participants who have received at least one dose of investigational product and have measurements of the respective endpoint at both baseline and Week 52.
Measure: Mean (Standard Deviation); unit: Percent A1C
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 140 | 179 | 173
Percent A1C | -0.68 (0.99) | -0.72 (0.95) | -0.96 (0.88)

13. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 52 (Excluding Rescue Therapy)
Description: Blood glucose was measured on a fasting basis. Blood was drawn at predose on Day 1 and after 52 weeks of treatment to determine change in plasma glucose levels (i.e., FPG at Week 52 minus FPG at Week 0). Participants who met pre-specified glycemic criteria were rescued with oral tablets of open-label glimepiride or basal insulin injected subcutaneously, and dosed according to Investigator judgment. Per protocol, this data set excludes data for any participant after the initiation of glycemic rescue therapy.
Time Frame: Baseline and Week 52
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 136 | 173 | 173
mg/dL | -12.0 (40.0) | -22.4 (39.3) | -35.2 (40.7)

14. Secondary Outcome: Percentage of Participants With an A1C of <7% (53 mmol/Mol) at Week 52 (Excluding Rescue Approach)
Description: as for outcome 6
Time Frame: Week 52
Population: All randomized participants who received at least one dose of investigational product. Any participant without post-baseline data at Week 52 was assumed to be "not at goal", where goal was A1C <7%, for the calculation of the percentages.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 209 | 207 | 205
Percentage of Participants | 30.6 | 34.8 | 36.6

15. Secondary Outcome: Percentage of Participants With an A1C of <6.5% (48 mmol/Mol) at Week 52 (Excluding Rescue Approach)
Description: A1C is blood marker used to report average blood glucose levels over prolonged periods of time. Percentage A1C is the ratio of glycated hemoglobin to total hemoglobin x 100. Participants who met pre-specified glycemic criteria were rescued with oral tablets of open-label glimepiride or basal insulin injected subcutaneously, and dosed according to Investigator judgment. Per protocol, this data set excludes data for any participant after the initiation of glycemic rescue therapy.
Time Frame: Week 52
Population: All randomized participants who received at least one dose of investigational product. Any participant without post-baseline data at Week 52 was assumed to be "not at goal", where goal was A1C <6.5%, for the calculation of the percentages.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 209 | 207 | 205
Percentage of Participants | 11.0 | 10.6 | 14.6

16. Secondary Outcome: Percentage of Participants Receiving Glycemic Rescue Therapy up to Week 52
Description: as for outcome 10
Time Frame: Up to Week 52
Population: All participants who received at least one dose of investigational product.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 209 | 207 | 205
Percentage of Participants | 17.2 [12.37 to 23.04] | 4.3 [2.01 to 8.09] | 1.5 [0.3 to 4.22]

17. Secondary Outcome: Change From Baseline in Body Weight at Week 52 (Excluding Rescue Approach)
Description: The change in body weight from baseline reflects the Week 52 body weight minus the Week 0 body weight. Participants who met pre-specified glycemic criteria were rescued with oral tablets of open-label glimepiride or basal insulin injected subcutaneously, and dosed according to Investigator judgment. Per protocol, this data set excludes data for any participant after the initiation of glycemic rescue therapy.
Time Frame: Baseline and Week 52
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 142 | 181 | 178
Kilograms | 0.07 (2.85) | -3.23 (3.68) | -3.35 (3.27)

18. Secondary Outcome: Change From Baseline in Sitting Systolic Blood Pressure at Week 52 (Excluding Rescue Approach)
Description: This change from baseline reflects the Week 52 sitting SBP minus the Week 0 sitting SBP. Participants who met pre-specified glycemic criteria were rescued with oral tablets of open-label glimepiride or basal insulin injected subcutaneously, and dosed according to Investigator judgment. Per protocol, this data set excludes data for any participant after the initiation of glycemic rescue therapy.
Time Frame: Baseline and Week 52
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 134 | 177 | 173
mmHg | 0.65 (13.38) | -2.63 (14.40) | -4.28 (13.28)

19. Secondary Outcome: Change From Baseline in Sitting Diastolic Blood Pressure at Week 52 (Excluding Rescue Approach)
Description: This change from baseline reflects the Week 52 sitting DBP minus the Week 0 sitting DBP. Participants who met pre-specified glycemic criteria were rescued with oral tablets of open-label glimepiride or basal insulin injected subcutaneously, and dosed according to Investigator judgment. Per protocol, this data set excludes data for any participant after the initiation of glycemic rescue therapy.
Time Frame: Baseline and Week 52
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 134 | 177 | 173
mmHg | 0.38 (8.16) | -1.40 (9.60) | -1.19 (7.74)

20. Secondary Outcome: Change From Baseline in A1C at Week 104 (Excluding Rescue Approach)
Description: A1C is blood marker used to report average blood glucose levels over prolonged periods of time. Percentage A1C is the ratio of glycated hemoglobin to total hemoglobin x 100. Thus, this change from baseline reflects the Week 104 A1C minus the Week 0 A1C. Participants who met pre-specified glycemic criteria were rescued with oral tablets of open-label glimepiride or basal insulin injected subcutaneously, and dosed according to Investigator judgment. Per protocol, this data set excludes data for any participant after the initiation of glycemic rescue therapy.
Time Frame: Baseline and Week 104
Population: All randomized participants who have received at least one dose of investigational product and have measurements of the respective endpoint at both baseline and Week 104.
Measure: Mean (Standard Deviation); unit: Percent A1C
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 109 | 147 | 142
Percent A1C | -0.58 (0.93) | -0.60 (0.97) | -0.89 (0.90)

21. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 104 (Excluding Rescue Approach)
Description: Blood glucose was measured on a fasting basis. Blood was drawn at predose on Day 1 and after 104 weeks of treatment to determine change in plasma glucose levels (i.e., FPG at Week 104 minus FPG at Week 0). Participants who met pre-specified glycemic criteria were rescued with oral tablets of open-label glimepiride or basal insulin injected subcutaneously, and dosed according to Investigator judgment. Per protocol, this data set excludes data for any participant after the initiation of glycemic rescue therapy.
Time Frame: Baseline and Week 104
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 104 | 143 | 144
mg/dL | -10.9 (44.3) | -18.2 (43.5) | -28.2 (44.9)

22. Secondary Outcome: Percentage of Participants With an A1C of <7% (53 mmol/Mol) at Week 104 (Excluding Rescue Approach)
Description: as for outcome 15
Time Frame: Week 104
Population: All randomized participants who received at least one dose of investigational product. Any participant without post-baseline data at Week 104 was assumed to be "not at goal", where goal was A1C <7%, for the calculation of the percentages.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 209 | 207 | 205
Percentage of Participants | 19.1 | 24.6 | 33.7

23. Secondary Outcome: Percentage of Participants With an A1C of <6.5% (48 mmol/Mol) at Week 104 (Excluding Rescue Approach)
Description: as for outcome 15
Time Frame: Week 104
Population: All randomized participants who received at least one dose of investigational product. Any participant without post-baseline data at Week 104 was assumed to be "not at goal", where goal was A1C <6.5% for the calculation of the percentages.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 209 | 207 | 205
Percentage of Participants | 7.2 | 10.6 | 12.2

24. Secondary Outcome: Percentage of Participants Receiving Glycemic Rescue Therapy up to Week 104
Description: Per protocol participants who met pre-specified glycemic criteria were rescued with oral tablets of open-label glimepiride or basal insulin injected subcutaneously, and dosed according to Investigator judgment.
Time Frame: Up to Week 104
Population: All participants who received at least one dose of investigational product.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 209 | 207 | 205
Percentage of participants | 24.4 [18.74 to 30.8] | 11.1 [7.18 to 16.2] | 10.7 [6.85 to 15.8]

25. Secondary Outcome: Change From Baseline in Body Weight at Week 104 (Excluding Rescue Approach)
Description: The change in body weight from baseline reflects the Week 104 body weight minus the Week 0 body weight. Participants who met pre-specified glycemic criteria were rescued with oral tablets of open-label glimepiride or basal insulin injected subcutaneously, and dosed according to Investigator judgment. Per protocol, this data set excludes data for any participant after the initiation of glycemic rescue therapy.
Time Frame: Baseline and Week 104
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 112 | 148 | 145
Kilograms | -0.18 (3.38) | -3.77 (4.29) | -3.63 (3.86)

26. Secondary Outcome: Change From Baseline in Sitting Systolic Blood Pressure at Week 104 (Excluding Rescue Approach)
Description: This change from baseline reflects the Week 104 sitting SBP minus the Week 0 sitting SBP. Participants who met pre-specified glycemic criteria were rescued with oral tablets of open-label glimepiride or basal insulin injected subcutaneously, and dosed according to Investigator judgment. Per protocol, this data set excludes data for any participant after the initiation of glycemic rescue therapy.
Time Frame: Baseline and Week 104
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 104 | 145 | 142
mmHg | 0.05 (13.76) | -3.61 (12.78) | -3.13 (14.11)

27. Secondary Outcome: Change From Baseline in Sitting Diastolic Blood Pressure at Week 104 (Excluding Rescue Approach)
Description: This change from baseline reflects the Week 104 sitting DBP minus the Week 0 sitting DBP. Participants who met pre-specified glycemic criteria were rescued with oral tablets of open-label glimepiride or basal insulin injected subcutaneously, and dosed according to Investigator judgment. Per protocol, this data set excludes data for any participant after the initiation of glycemic rescue therapy.
Time Frame: Baseline and Week 104
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 104 | 145 | 142
mmHg | -0.46 (8.77) | -2.36 (9.23) | -1.52 (8.61)

28. Secondary Outcome: Ertugliflozin Plasma Concentrations (ng/mL): Summary Statistics Over Time (Excluding Rescue Approach)
Description: Pharmacokinetic samples were collected at approximately 24 hours following the prior day's dose and before administration of the current day's dose. The lower limit of quantitation (LLOQ) was 0.500 mg/mL. Participants who met pre-specified glycemic criteria were rescued with oral tablets of open-label glimepiride or basal insulin injected subcutaneously, and dosed according to Investigator judgment. Per protocol, this data set excludes data for any participant after the initiation of glycemic rescue therapy.
Time Frame: Pre-dose and/or 60 minutes post-dose on Weeks 6, 12, 18, and 30
Population: All subjects as treated (including those with all concentrations below the lower limit of quantification) were included in the calculation of the summary statistics. Numbers of participants with non-missing concentrations at the respective time points are displayed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 209 | 207 | 205
ng/mL
  Week 6:Pre-dose: number analyzed (Participants) | 127 | 194 | 191
  Week 6:Pre-dose | NA (NA) — Below the lower limit of quantification | 14.89 (28.11) | 38.38 (74.83)
  Week 12:Pre-dose: number analyzed (Participants) | 125 | 196 | 186
  Week 12:Pre-dose | NA (NA) — Below the lower limit of quantification | 12.34 (26.07) | 29.23 (55.63)
  Week 12:60 mins post-dose: number analyzed (Participants) | 124 | 191 | 179
  Week 12:60 mins post-dose | NA (NA) — Below the lower limit of quantification | 74.84 (51.58) | 228.13 (139.14)
  Week 18:Pre-dose: number analyzed (Participants) | 110 | 202 | 190
  Week 18:Pre-dose | 0.01 (0.10) | 9.91 (21.18) | 24.46 (39.97)
  Week 18:60 mins post-dose: number analyzed (Participants) | 108 | 198 | 183
  Week 18:60 mins post-dose | 0.01 (0.09) | 74.39 (49.77) | 214.96 (147.36)
  Week 30:Pre-dose: number analyzed (Participants) | 52 | 196 | 187
  Week 30:Pre-dose | 0.15 (1.07) | 12.66 (25.50) | 30.55 (60.33)

29. Secondary Outcome: Percent Change From Baseline in BMD at Week 26 as Measured by DXA at the Lumbar Spine (L1-L4) Using Raw Data (Excluding Bone Rescue Approach)
Description: BMD at the femoral neck was assessed by DXA at Week 0 and Week 26. Participants who exhibited a significant reduction in BMD according to the protocol defined criteria completed an unscheduled DXA scan and, if required, received bone-active therapy. This table excludes measurements obtained after initiation of bone rescue medications.
Time Frame: Baseline and Week 26
Population: All randomized participants who have received at least one dose of investigational product and have a measurement at baseline and at least one post-baseline measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 191 | 200 | 189
Percentage change | 0.22 [-0.20 to 0.65] | -0.01 [-0.42 to 0.41] | 0.12 [-0.31 to 0.55]
Statistical Analysis 1: Comparison: Placebo/Glimepiride vs Ertugliflozin 15 mg; Test type: Other; Difference in the Least Squares Means = -0.10, 95% CI 2-sided [-0.71 to 0.50]; Based on cLDA model with fixed effects for treatment, time, prior antihyperglycemic medication (Metformin monotherapy or Metformin + another AHA), baseline eGFR (continuous), menopausal status, and the interaction of time by treatment. Time was treated as a categorical variable
Statistical Analysis 2: Comparison: Placebo/Glimepiride vs Ertugliflozin 5 mg; Test type: Other; Difference in the Least Squares Means = -0.23, 97% CI 2-sided [-0.83 to 0.37]; [other analysis details as in outcome 29, analysis 1]

30. Secondary Outcome: Percent Change From Baseline in BMD at Week 26 as Measured by DXA at the Femoral Neck Using Raw Data (Excluding Bone Rescue Approach)
Description: as for outcome 29
Time Frame: Baseline and Week 26
Population: as for outcome 29
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 191 | 200 | 190
Percent change | -0.40 [-0.89 to 0.09] | -0.10 [-0.57 to 0.38] | 0.30 [-0.19 to 0.79]
Statistical Analysis 1: Comparison: Placebo/Glimepiride vs Ertugliflozin 15 mg; Test type: Other; Difference in the Least Squares Means = 0.70, 95% CI 2-sided [0.00 to 1.39]; [other analysis details as in outcome 29, analysis 1]
Statistical Analysis 2: Comparison: Placebo/Glimepiride vs Ertugliflozin 5 mg; Test type: Other; Difference in the Least Squares Means = 0.30, 95% CI 2-sided [-0.38 to 0.99]; [other analysis details as in outcome 29, analysis 1]

31. Secondary Outcome: Percent Change From Baseline in BMD at Week 26 as Measured by DXA at the Total Hip Using Raw Data (Excluding Bone Rescue Approach)
Description: BMD at the total hip was assessed by DXA at Week 0 and Week 26. Participants who exhibited a significant reduction in BMD according to the protocol defined criteria completed an unscheduled DXA scan and, if required, received bone-active therapy. This table excludes measurements obtained after initiation of bone rescue medications.
Time Frame: Baseline and Week 26
Population: as for outcome 29
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 191 | 200 | 190
Percent change | -0.63 [-0.92 to -0.34] | -0.55 [-0.83 to -0.27] | -0.36 [-0.65 to -0.07]
Statistical Analysis 1: Comparison: Placebo/Glimepiride vs Ertugliflozin 15 mg; Test type: Other; Difference in the Least Squares Means = 0.27, 95% CI 2-sided [-0.15 to 0.68]; [other analysis details as in outcome 29, analysis 1]
Statistical Analysis 2: Comparison: Placebo/Glimepiride vs Ertugliflozin 5 mg; Test type: Other; Difference in the Least Squares Means = 0.08, 95% CI 2-sided [-0.33 to 0.48]; [other analysis details as in outcome 29, analysis 1]

32. Secondary Outcome: Percent Change From Baseline in BMD at Week 26 as Measured by DXA at the Distal Forearm Using Raw Data (Excluding Bone Rescue Approach)
Description: BMD at the distal forearm was assessed by DXA at Week 0 and Week 26. Participants who exhibited a significant reduction in BMD according to the protocol defined criteria completed an unscheduled DXA scan and, if required, received bone-active therapy. This table excludes measurements obtained after initiation of bone rescue medications.
Time Frame: Baseline and Week 26
Population: as for outcome 29
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 190 | 200 | 189
Percent change | 0.06 [-0.35 to 0.47] | -0.15 [-0.55 to 0.24] | -0.13 [-0.53 to 0.28]
Statistical Analysis 1: Comparison: Placebo/Glimepiride vs Ertugliflozin 15 mg; Test type: Other; Difference in the Least Squares Means = -0.19, 95% CI 2-sided [-0.76 to 0.39]; Based on cLDA model with fixed effects for treatment, time, prior anti hyperglycemic medication (Metformin monotherapy or Metformin + another AHA), baseline eGFR (continuous), menopausal status, and the interaction of time by treatment. Time was treated as a categorical variable
Statistical Analysis 2: Comparison: Placebo/Glimepiride vs Ertugliflozin 5 mg; Test type: Other; Difference in the Least Squares Means = -0.21, 95% CI 2-sided [-0.78 to 0.35]; [other analysis details as in outcome 32, analysis 1]

33. Secondary Outcome: Percent Change From Baseline in Bone Biomarker Carboxy-Terminal Cross-Linking Telopeptides of Type I Collagen (CTX) at Week 26 (Excluding Bone Rescue Approach)
Description: CTX is a biochemical marker of bone resorption. Participants who exhibited a significant reduction in BMD according to the protocol defined criteria completed an unscheduled DXA scan and, if required, received bone-active therapy. This table excludes measurements obtained after initiation of bone rescue medications.
Time Frame: Baseline and Week 26
Population: All randomized participants who have received at least one dose of investigational product and have measurements of the respective endpoint at both baseline and Week 26.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 185 | 179 | 180
Percent change | 10.8 (106.6) | 51.9 (121.9) | 80.2 (149.7)

34. Secondary Outcome: Percent Change From Baseline in Bone Biomarker Procollagen Type I N-terminal Propeptide (P1NP) at Week 26 (Excluding Bone Rescue Approach)
Description: P1NP is a biochemical marker of bone resorption. Participants who exhibited a significant reduction in BMD according to the protocol defined criteria completed an unscheduled DXA scan and, if required, received bone-active therapy. This table excludes measurements obtained after initiation of bone rescue medications.
Time Frame: Baseline and Week 26
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 186 | 183 | 183
Percent change | 0.5 (11.7) | 0.8 (12.1) | 0.5 (15.0)

35. Secondary Outcome: Percent Change From Baseline in Bone Biomarker Parathyroid Hormone (PTH) at Week 26 (Excluding Bone Rescue Approach)
Description: PTH is a biochemical marker of bone resorption. Participants who exhibited a significant reduction in BMD according to the protocol defined criteria completed an unscheduled DXA scan and, if required, received bone-active therapy. This table excludes measurements obtained after initiation of bone rescue medications.
Time Frame: Baseline and Week 26
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 186 | 182 | 184
Percent change | -0.98 (6.71) | 0.28 (7.52) | 0.14 (7.53)

36. Secondary Outcome: Percent Change From Baseline in BMD at Week 52 as Measured by DXA at the Lumbar Spine (L1-L4) Using Raw Data (Excluding Bone Rescue Approach)
Description: BMD at the femoral neck was assessed by DXA at Week 0 and Week 52. Participants who exhibited a significant reduction in BMD according to the protocol defined criteria completed an unscheduled DXA scan and, if required, received bone-active therapy. This table excludes measurements obtained after initiation of bone rescue medications.
Time Frame: Baseline and Week 52
Population: as for outcome 29
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 191 | 202 | 189
Percent change | -0.10 [-0.60 to 0.40] | -0.28 [-0.77 to 0.20] | 0.07 [-0.43 to 0.57]
Statistical Analysis 1: Comparison: Placebo/Glimepiride vs Ertugliflozin 15 mg; Test type: Other; Difference in the Least Squares Means = 0.17, 95% CI 2-sided [-0.53 to 0.88]; [other analysis details as in outcome 29, analysis 1]
Statistical Analysis 2: Comparison: Placebo/Glimepiride vs Ertugliflozin 5 mg; Test type: Other; Difference in the Least Squares Means = -0.18, 97% CI 2-sided [-0.88 to 0.51]; [other analysis details as in outcome 29, analysis 1]

37. Secondary Outcome: Percent Change From Baseline in BMD at Week 52 as Measured by DXA at the Femoral Neck Using Raw Data (Excluding Bone Rescue Approach)
Description: as for outcome 36
Time Frame: Baseline and Week 52
Population: as for outcome 29
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 191 | 202 | 190
Percent change | -0.69 [-1.25 to -0.14] | -0.49 [-1.04 to 0.06] | -0.44 [-1.06 to 0.17]
Statistical Analysis 1: Comparison: Placebo/Glimepiride vs Ertugliflozin 15 mg; Test type: Other; Difference in the Least Squares Means = 0.25, 95% CI 2-sided [-0.48 to 0.98]; [other analysis details as in outcome 29, analysis 1]
Statistical Analysis 2: Comparison: Placebo/Glimepiride vs Ertugliflozin 5 mg; Test type: Other; Difference in the Least Squares Means = 0.20, 95% CI 2-sided [-0.51 to 0.91]; [other analysis details as in outcome 29, analysis 1]

38. Secondary Outcome: Percent Change From Baseline in BMD at Week 52 as Measured by DXA at the Total Hip Using Raw Data (Excluding Bone Rescue Approach)
Description: BMD at the total hip was assessed by DXA at Week 0 and Week 52. Participants who exhibited a significant reduction in BMD according to the protocol defined criteria completed an unscheduled DXA scan and, if required, received bone-active therapy. This table excludes measurements obtained after initiation of bone rescue medications.
Time Frame: Baseline and Week 52
Population: as for outcome 29
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 191 | 202 | 190
Percent change | -0.82 [-1.19 to -0.46] | -1.04 [-1.41 to -0.67] | -1.32 [-1.69 to -0.94]
Statistical Analysis 1: Comparison: Placebo/Glimepiride vs Ertugliflozin 15 mg; Test type: Other; Difference in the Least Squares Means = -0.50, 95% CI 2-sided [-0.95 to -0.04]; [other analysis details as in outcome 29, analysis 1]
Statistical Analysis 2: Comparison: Placebo/Glimepiride vs Ertugliflozin 5 mg; Test type: Other; Difference in the Least Squares Means = -0.22, 95% CI 2-sided [-0.66 to 0.23]; [other analysis details as in outcome 29, analysis 1]

39. Secondary Outcome: Percent Change From Baseline in BMD at Week 52 as Measured by DXA at the Distal Forearm Using Raw Data (Excluding Bone Rescue Approach)
Description: BMD at the distal forearm was assessed by DXA at Week 0 and Week 52. Participants who exhibited a significant reduction in BMD according to the protocol defined criteria completed an unscheduled DXA scan and, if required, received bone-active therapy. This table excludes measurements obtained after initiation of bone rescue medications.
Time Frame: Baseline and Week 52
Population: as for outcome 29
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 190 | 200 | 189
Percent change | -0.44 [-0.95 to 0.06] | -0.59 [-1.04 to 0.14] | -0.39 [-0.90 to 0.12]
Statistical Analysis 1: Comparison: Placebo/Glimepiride vs Ertugliflozin 15 mg; Test type: Other; Difference in the Least Squares Means = 0.06, 95% CI 2-sided [-0.61 to 0.72]; [other analysis details as in outcome 32, analysis 1]
Statistical Analysis 2: Comparison: Placebo/Glimepiride vs Ertugliflozin 5 mg; Test type: Other; Difference in the Least Squares Means = -0.15, 95% CI 2-sided [-0.78 to 0.49]; [other analysis details as in outcome 32, analysis 1]

40. Secondary Outcome: Percent Change From Baseline in Bone Biomarker CTX at Week 52 (Excluding Bone Rescue Approach)
Description: as for outcome 33
Time Frame: Baseline and Week 52
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 171 | 178 | 171
Percent change | 15.54 (43.34) | 34.36 (52.74) | 41.57 (50.69)

41. Secondary Outcome: Percent Change From Baseline in Bone Biomarker P1NP at Week 52 (Excluding Bone Rescue Approach)
Description: as for outcome 34
Time Frame: Baseline and Week 52
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 171 | 179 | 173
Percent Change | 24.50 (120.29) | 8.41 (30.95) | 19.79 (79.57)

42. Secondary Outcome: Percent Change From Baseline in Bone Biomarker PTH at Week 52 (Excluding Bone Rescue Approach)
Description: as for outcome 35
Time Frame: Baseline and Week 52
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 171 | 177 | 175
Percent Change | 8.11 (52.05) | 11.09 (41.80) | 2.48 (36.57)

43. Secondary Outcome: Percent Change From Baseline in BMD at Week 104 as Measured by DXA at the Lumbar Spine (L1-L4) Using Raw Data (Excluding Bone Rescue Approach)
Description: BMD at the femoral neck was assessed by DXA at Week 0 and Week 104. Participants who exhibited a significant reduction in BMD according to the protocol defined criteria completed an unscheduled DXA scan and, if required, received bone-active therapy. This table excludes measurements obtained after initiation of bone rescue medications.
Time Frame: Baseline and Week 104
Population: as for outcome 29
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 191 | 202 | 189
Percent change | 0.09 [-0.47 to 0.66] | -0.19 [-0.72 to 0.35] | -0.13 [-0.68 to 0.42]
Statistical Analysis 1: Comparison: Placebo/Glimepiride vs Ertugliflozin 15 mg; Test type: Other; Difference in the Least Squares Means = -0.23, 95% CI 2-sided [-1.01 to 0.56]; [other analysis details as in outcome 29, analysis 1]
Statistical Analysis 2: Comparison: Placebo/Glimepiride vs Ertugliflozin 5 mg; Test type: Other; Difference in the Least Squares Means = -0.28, 97% CI 2-sided [-1.06 to 0.50]; [other analysis details as in outcome 29, analysis 1]

44. Secondary Outcome: Percent Change From Baseline in BMD at Week 104 as Measured by DXA at the Femoral Neck Using Raw Data (Excluding Bone Rescue Approach)
Description: as for outcome 43
Time Frame: Baseline and Week 104
Population: as for outcome 29
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 191 | 202 | 190
Percent change | -1.23 [-1.86 to -0.61] | -1.11 [-1.74 to -0.49] | -0.96 [-1.67 to -0.26]
Statistical Analysis 1: Comparison: Placebo/Glimepiride vs Ertugliflozin 15 mg; Test type: Other; Difference in the Least Squares Means = 0.27, 95% CI 2-sided [-0.58 to 1.13]; [other analysis details as in outcome 29, analysis 1]
Statistical Analysis 2: Comparison: Placebo/Glimepiride vs Ertugliflozin 5 mg; Test type: Other; Difference in the Least Squares Means = 0.12, 95% CI 2-sided [-0.70 to 0.93]; [other analysis details as in outcome 29, analysis 1]

45. Secondary Outcome: Percent Change From Baseline in BMD at Week 104 as Measured by DXA at the Total Hip Using Raw Data (Excluding Bone Rescue Approach)
Description: BMD at the total hip was assessed by DXA at Week 0 and Week 104. Participants who exhibited a significant reduction in BMD according to the protocol defined criteria completed an unscheduled DXA scan and, if required, received bone-active therapy. This table excludes measurements obtained after initiation of bone rescue medications.
Time Frame: Baseline and Week 104
Population: as for outcome 29
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 191 | 202 | 190
Percent change | -1.18 [-1.63 to -0.73] | -1.72 [-2.19 to -1.25] | -2.02 [-2.51 to -1.53]
Statistical Analysis 1: Comparison: Placebo/Glimepiride vs Ertugliflozin 15 mg; Test type: Other; Difference in the Least Squares Means = -0.84, 95% CI 2-sided [-1.44 to -0.24]; [other analysis details as in outcome 29, analysis 1]
Statistical Analysis 2: Comparison: Placebo/Glimepiride vs Ertugliflozin 5 mg; Test type: Other; Difference in the least Squares Means = -0.54, 95% CI 2-sided [-1.12 to 0.05]; [other analysis details as in outcome 29, analysis 1]

46. Secondary Outcome: Percent Change From BMD at Week 104 as Measured by DXA at the Distal Forearm Using Raw Data (Excluding Bone Rescue Approach)
Description: BMD at the distal forearm was assessed by DXA at Week 0 and Week 104. Participants who exhibited a significant reduction in BMD according to the protocol defined criteria completed an unscheduled DXA scan and, if required, received bone-active therapy. This table excludes measurements obtained after initiation of bone rescue medications.
Time Frame: Baseline and Week 104
Population: as for outcome 29
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 190 | 200 | 189
Percent change | -0.58 [-1.13 to -0.03] | -0.40 [-0.87 to 0.06] | -0.64 [-1.19 to -0.09]
Statistical Analysis 1: Comparison: Placebo/Glimepiride vs Ertugliflozin 15 mg; Test type: Other; Difference in the Least Squares Means = -0.06, 95% CI 2-sided [-0.77 to 0.65]; [other analysis details as in outcome 32, analysis 1]
Statistical Analysis 2: Comparison: Placebo/Glimepiride vs Ertugliflozin 5 mg; Test type: Other; Difference in the Least Squares Means = 0.18, 95% CI 2-sided [-0.50 to 0.85]; [other analysis details as in outcome 32, analysis 1]

47. Secondary Outcome: Percent Change From Baseline in Bone Biomarker CTX at Week 104 (Excluding Bone Rescue Approach)
Description: as for outcome 33
Time Frame: Baseline and Week 104
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 149 | 160 | 159
Percent change | 19.29 (71.73) | 26.94 (58.44) | 32.53 (59.29)

48. Secondary Outcome: Percent Change From Baseline in Bone Biomarker P1NP at Week 104 (Excluding Bone Rescue Approach)
Description: as for outcome 34
Time Frame: Baseline and Week 104
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 149 | 162 | 162
Percent change | 19.38 (93.02) | 10.11 (39.14) | 24.21 (83.23)

49. Secondary Outcome: Percent Change From Baseline in Bone Biomarker PTH at Week 104 (Excluding Bone Rescue Approach)
Description: as for outcome 35
Time Frame: Baseline and Week 104
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
Number analyzed (Participants) | 148 | 158 | 161
Percent change | 10.12 (60.13) | 8.16 (40.97) | 5.46 (38.53)

ADVERSE EVENTS:
Time Frame: Up to 106 weeks
Description: Participants who met pre-specified glycemic criteria were rescued with open-label glimepiride or insulin glargine according to Investigator judgment. The analysis population was all participants who received at least one dose of investigational product. Adverse events were reported for the all post-randomization follow-up period.
Arm/Group | Placebo/Glimepiride | Ertugliflozin 5 mg | Ertugliflozin 15 mg
All-Cause Mortality (participants affected / at risk) | 3/209 | 1/207 | 2/205
Serious Adverse Events (participants affected / at risk) | 22/209 | 20/207 | 20/205
Other Adverse Events (participants affected / at risk) | 103/209 | 79/207 | 100/205
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/Glimepiride (N=209) | Ertugliflozin 5 mg (N=207) | Ertugliflozin 15 mg (N=205)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 1 (2)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial bridging (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Cardiac death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Osteomyelitis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Otitis media chronic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Limb crushing injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Necrotising myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/Glimepiride (N=209) | Ertugliflozin 5 mg (N=207) | Ertugliflozin 15 mg (N=205)
Influenza (Infections and infestations) | 12 (13) | 11 (13) | 10 (13)
Upper respiratory tract infection (Infections and infestations) | 33 (44) | 23 (30) | 21 (22)
Urinary tract infection (Infections and infestations) | 13 (18) | 6 (9) | 17 (22)
Viral upper respiratory tract infection (Infections and infestations) | 21 (27) | 12 (16) | 9 (11)
Weight decreased (Investigations) | 3 (3) | 9 (9) | 15 (15)
Hypoglycaemia (Metabolism and nutrition disorders) | 43 (213) | 14 (119) | 18 (66)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 7 (9) | 11 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 9 (10) | 20 (20)
Headache (Nervous system disorders) | 10 (15) | 14 (18) | 11 (15)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 8 (8) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator will provide manuscripts, abstracts, or the full text of any other intended disclosure (poster presentation, invited speaker or guest lecturer presentation, etc.) to the Sponsor at least 30 days before they are submitted for publication or otherwise disclosed. If any patent action is required to protect intellectual property rights, Investigator agrees to delay the disclosure for a period not to exceed an additional 60 days.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-09-20): https://cdn.clinicaltrials.gov/large-docs/89/NCT02033889/Prot_SAP_000.pdf